CLINICAL TRIAL: NCT02564562
Title: A Phase 1 Open-Label, Radiolabeled, Single-Dose Study To Investigate The Absorption, Distribution, Metabolism, And Excretion Of [14c]PF-06463922 In Healthy Male Volunteers
Brief Title: A Study To Investigate The Absorption, Distribution, Metabolism, And Excretion Of [14c]PF-06463922 In Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: B7461004
Record Dates: First submitted 2015-09-29; First posted 2015-09-30 (Estimated); Last update posted 2015-12-04 (Estimated); Status verified 2015-12

CONDITIONS: Healthy
Keywords: PF-06463922; [14C]PF-06463922; Human ADME; Radiolabel; Mass Balance; Pharmacokinetics
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (Experimental): Radiolabeled PF-06463922 in healthy volunteers
  Interventions: Drug: [14C] PF-06463922

INTERVENTIONS:
Drug: [14C] PF-06463922 — Single oral dose of 100mg PF-06463922 + [14C] PF-06463922

SUMMARY:
The study aims to understand, using radiolabelled PF-06463922, how this compound is modified by the body once it is absorbed. The study also aims to understand how much of the compound is broken down and how much leaves the body unchanged.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects who, at the time of screening, are between the ages of 18 and 55 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 30.5 kg/m2 and a total body weight >50 kg (110 lbs)
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study.
* Subjects who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy).
* A positive urine drug screen.
* History of regular alcohol consumption exceeding 7 drinks/week (1 drink = 5 ounces [150 mL] of wine or 12 ounces [360 mL] of beer or 1.5 ounces [45 mL] of hard liquor) within 6 months of Screening.
* Treatment with an investigational drug within 30 days (or as determined by the local requirement) or 5 half-lives preceding the first dose of study medication (whichever is longer).
* Screening supine blood pressure 140 mm Hg (systolic) or 90 mm Hg (diastolic), following at least 5 minutes of supine rest. If blood pressure is 140 mm Hg (systolic) or 90 mm Hg (diastolic), the blood pressure should be repeated two more times and the average of the three blood pressure values should be used to determine the subject's eligibility.
* Screening supine 12-lead ECG demonstrating QTcF (time from ECG Q wave to the end of the T wave corresponding to electrical systole [QT] corrected for the heart rate using the Fredericia's formula) >450 msec or a QRS interval (time from ECG Q wave to the end of the S wave corresponding to ventricle depolarization) >120 msec. If QTcF exceeds 450 msec, or QRS exceeds 120 msec, the ECG should be repeated two more times and the average of the three QTcF or QRS values should be used to determine the subject's eligibility.
* Subjects with ANY of the following abnormalities in clinical laboratory tests at screening, as assessed by the study specific laboratory and confirmed by a single repeat, if deemed necessary:

  * Aspartate aminotransferase (AST)/serum glutamic oxaloacetic transminase (SGOT) or alanine aminotransferase (ALT)/serum glutamic pyruvic transminase (SGPT) 3 x upper limit of normal (ULN);
  * Total bilirubin ≥ 1.5x ULN; subjects with a history of Gilbert's syndrome may have a direct bilirubin measured and would be eligible for this study provided the direct bilirubin is ≤ ULN.
* Use of prescription or nonprescription drugs and dietary supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of study medication. As an exception, acetaminophen/paracetamol may be used at doses of 1 g/day. Limited use of non-prescription medications that are not believed to affect subject safety or the overall results of the study may be permitted on a case-by-case basis following approval by the sponsor.

Herbal supplements and hormone replacement therapy must be discontinued at least 28 days prior to the first dose of study medication.

* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 56 days prior to dosing.
* History of sensitivity to heparin or heparin-induced thrombocytopenia.
* Unwilling or unable to comply with the Lifestyle guidelines described in this protocol.
* Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the conduct of the study.
* Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.
* Subjects with a history of irregular bowel movements eg, regular episodes of diarrhea or constipation, irritable bowel syndrome (IBS) or lactose intolerance.
* Subjects enrolled in a previous radionucleotide study or who have received radiotherapy within 12 months prior to screening or such that total radioactivity would exceed acceptable dosimetry (ie, occupational exposure of 5 rem per year).
* Subjects whose occupation requires exposure to radiation or monitoring of radiation exposure.
* Subjects who have used tobacco within 90 days prior to dosing.
* Male subjects with partners currently pregnant; male subjects able to father children who are unwilling or unable to use 2 highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 90 days after the last dose of investigational product or longer based upon the compound's half life characteristics.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2015-10; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Mass Balance | 14 days
  Mass balance: Cumulative recovery (%) of total radioactivity in urine and feces.
Metabolic profiling / metabolite identification in plasma, urine, and fecal samples | 14 days
AUCinf | 14 days
  Area Under the Curve From Time Zero to Extrapolated Infinite Time
AUClast | 14 days
  Area under the plasma concentration time profile from time 0 to the time of the last quantifiable concentration (Clast)
kel | 14 days
  Elimination rate constant
Cmax | 14 days
  Maximum observed plasma concentration
Tmax | 14 days
  Time for Cmax
t1/2 | 14 days
  Terminal elimination half life
CL/F | 14 days
  Apparent oral clearance
Ae | 14 days
  Total amount of unchanged drug excreted in the urine from time 0 to discharge day
Ae% | 14 days
  Total amount of unchanged drug excreted in the urine from time 0 to infinity expressed as percent of dose
Clr | 14 days
  Renal Clearance
Crbc | 14 days
  Total radioactivity in RBCs
Vz/F | 14 days
  Apparent volume of distribution following oral administration

SECONDARY OUTCOMES:
AUC (0-24) | 14 days
  Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0 - 24). It is obtained from AUC (0 - t) plus AUC (t - 24).

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Covance Clinical Research Unit Inc., Madison, Wisconsin, United States